CLINICAL TRIAL: NCT02547467
Title: Epidemiological Survey of Death Modalities in Patients With Septic Shock Referred to French Intensive Care Units: TOADS Study.
Brief Title: TOADS Study: TO Assess Death From Septic Shock.
Acronym: TOADS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: 49RC14_0223
Record Dates: First submitted 2015-07-08; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Septic Shock
Keywords: mortality
MeSH Terms: conditions — Shock, Septic | interventions — Epidemiologic Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: epidemiologic study — There is no intervention as it is a pure observational study for epidemiologic survey.

SUMMARY:
The aim of this study is to assess the causes of death in patients with septic shock in French intensive care units. It is an epidemiologic and descriptive study .

DETAILED DESCRIPTION:
The purpose of this epidemiologic study is to describe with accuracy the reasons and causes of death in patients with septic shock during patients stay in intensive care units. All deceased patients with primary diagnosis of septic shock will be included in this survey and patients baseline characteristics as well as the clinical and data at the time of patient's death will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Died of septic shock in the intensive care unit (ICU)
* At least 6 hours of vasopressors

Exclusion Criteria:

* Legally protected adult patient.
* Less than 6 hours of vasopressors
* Opposition to participation in the study expressed by the patient, family or person of trust

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who had died of septic shock
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study is to identify the reasons of death of patients with septic shock via a questionnaire. | Patients will be followed during their hospital stay, with a maximal follow up of 90 days
  Recording of the context and the cause of death with a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ASFAR, MD-PhD, Study Director — University hospital, Angers, FRANCE